CLINICAL TRIAL: NCT05952921
Title: Hypochlorous Acid as a Potential Postsurgical Antimicrobial Agent in Periodontitis. A Non-inferiority Randomized Controlled Trial.
Brief Title: Comparison of the Effectiveness of Hypochlorous Acid and Chlorhexidine as a Post-surgical Antimicrobial Agent
Acronym: HOCl-Post-AA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, David Díaz-Báez, Clinical Professor, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UnBosque-HOCl-003
Record Dates: First submitted 2023-06-30; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Diseases; Chronic Periodontitis; Microbial Colonization
Keywords: Chlorhexidine; HOCl; bacterial recolonization; antiplaque
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis; Communicable Diseases | interventions — Mouthwashes; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The rinses will be coded to avoid any bias and the codes will not be broken before the study ends. Patients will be randomly assigned to receive a rinse bottle identified as solution "A" or "B". These bottles will be identical in terms of shape, color and material. Neither the subject nor the dentists will be informed about the group assignment. The principal investigator who does not participate in the treatment or data collection will have access to a closed envelope with the allocation information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypochlorous acid (Experimental): Thirty-two voluntary participants were randomly assigned to receive one of two post-surgical protocols after periodontal surgery: a high concentration rinse with 0.05% HOCl (7 days), followed by 0.025% HOCl /(14 days)
  Interventions: Other: Mouthwash
- Chlorhexidine (Active Comparator): Thirty-two voluntary participants were randomly assigned to receive one of two post-surgical protocols after periodontal surgery: a high concentration of 0.2% CHX (7 days), followed by 0.012% CHX (14 days).
  Interventions: Other: Chlorhexidine

INTERVENTIONS:
Other: Mouthwash — Concentration rinse with 0.05% HOCl
  Arms: Hypochlorous acid
Other: Chlorhexidine — A high concentration of 0.2% CHX (7 days), followed by 0.012% CHX (14 days).
  Arms: Chlorhexidine

SUMMARY:
The aim of the study is to evaluate the effectiveness of Hypochlorous Acid and Chlorhexidine as postsurgical antimicrobial agents in the treatment of severe chronic periodontal disease. The selected patients will be randomly divided into two groups of 16 each. Subjects in group I will undergo scaling and surgical root planing and will use mouthrinse with 0.05% HOCl for 7 days, after this they will mouthwash with 0.025% HOCl until day 21 and Subjects in group II will undergo scaling and surgical root planing followed by a rinse with CHX 0.2% for 7 days, after this they will mouthwash with 0.12% CHX until day 21. Null Hypothesis: There are no significant differences between hypochlorous acid and chlorhexidine in reducing plaque formation at 7, 21 and 90 days of evaluation.

There are no significant differences between HOCl and CHX in the elimination or reduction of periodontopathogenic microorganisms at 7, 21 and 90 days. Alternative hypotheses: There are significant differences between hypochlorous acid and chlorhexidine in reducing plaque formation at 7, 21 and 90 days of evaluation. There are significant differences between HOCl and CHX in the elimination or reduction of periodontopathogenic microorganisms at 7, 21 and 90 days.

DETAILED DESCRIPTION:
For the HOCl effectiveness study, parallel groups were compared to determine the clinical and microbiological effectiveness of hypochlorous acid by evaluating the reduction of plaque index, gingival index and clinical insertion level as a primary outcome with chlorhexidine, for a period of 7, 21 and 90 days. The selected patients will be randomly divided into two groups of 16 each. Subjects in group I: 16 subjects for scaling and surgical root planing (surgical technique Modified Widman) and HOCl 0.05% for 7 days and HOCl 0.025% until day 21 and Subjects in group II: 16 subjects for scaling and surgical root planing (surgical technique Modified Widman) and CHX 0.2% for 7 days and 0.12% CHX until day 21. At the beginning of the study (day0) all patients will be evaluated the plaque index, gingival index, periodontal chart, saliva sample collection and subgingival microbiological test, all will receive surgical periodontal treatment (scaling and surgical root planing surgical technique Modified Widman) after the surgery will be instructed to rinse with 15 ml twice a day for 30 seconds in the morning 30 minutes after breakfast and brushing teeth, and at night, before going to sleep with one of the two Rinses: HOCl 0.05% for the first seven days and 0.025% from day eight to day 21 and CHX 0.2% for the first seven days and 0.12% from day eight to day 21. The rinses were coded to avoid any bias and the codes will not be broken before the study ends. Patients will be assigned randomly each will receive a flushing flask identified as solution "A" or "B". These bottles will be identical in terms of shape, color and material. Neither the subject nor the dentists will be informed about the group assignment. The principal investigator who does not participate in the treatment or data collection will have access to a closed envelope with the allocation information. Each of the participants will be clear that the area where the surgical procedure should be performed should remain unbrushed for 21 days. After 21 days all individuals will be given a special toothbrush for after surgery and indications are given for the brushing of the operated area. Adverse effects were evaluated both microbiologically to verify the absence or presence of opportunistic flora associated with the use of mouthwashes and effects on teeth and mucous membranes using a survey and clinical assessment.

The data will be collected as follows:

Day zero will evaluate plaque and gingival index, periodontal pocket depth al probing, clinical insertion level, saliva uptake and subgingival sampling for microbiological analysis. On day 7 suture removal and plaque and gingival index, saliva sampling and subgingival sampling for microbiological analysis were evaluated. On day 21, plaque and gingival index, saliva sampling and subgingival sampling will be evaluated for microbiological analysis. And on day 90, plaque and gingival index, periodontal pocket depth at probing, clinical insertion level, saliva sampling and subgingival sampling for microbiological analysis.

For the test the following parameters will be evaluated: Gingival Index and Plaque Index. The modified gingival index and the modified visible plaque index will be evaluated. Four evaluations will be performed: one at the beginning of the study, another at day 7, 21 and the last at day 90 and the Index of visible plaque and Gingival index (Modified Silness & Loe) will be used. The probing depth and the level of clinical insertion will be measured in six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual and mesiolingual) exclusion of the third molar, on day 0 and 90. Measurements will be recorded in the periodontal chart and a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) will be used. Sampling of saliva and microbial count: Microbiological samples in saliva and subgingival will be collected before surgery (day 0) and after surgery at day 7, 21 and 90. For the sampling of subgingival bacteria, the selected sites were cleaned (sterile curettes) before sampling, with cotton roll the field is isolated and dried carefully to avoid contamination, bacterial samples will be collected with paper tips of endodontics sterile (size 55 absorbent paper, Dentsply, Maillefer). Samples will be individually placed in labeled Eppendorf tubes containing Buffer, kept at -70°C and then sent to the laboratory. Will be processed in the laboratory of Oral Microbiology of the Universidad el Bosque. Samples will be analyzed using the real-time PCR technique.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Age between 20 and 60 years.
* Diagnosis of chronic periodontitis.
* Minimum 20 teeth and minimum 3 teeth with at least one site with PD≥5 mm and CAL> 4 mm
* Radiographic evidence of bone loss.
* Good general health.

Exclusion Criteria:

* Prior periodontal therapy.
* Smokers.
* Antibiotic therapy in the last 4 months, consumption of NSAIDs.
* Pregnancy and / or breastfeeding.
* Systemic pathology that may affect the progression of PD.
* Allergy to HOCl or CHX.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) | Baseline
  Presence or absence of visible plaque evaluated with a periodontal probe
Plaque Index (PI) | 7 days
  Presence or absence of visible plaque evaluated with a periodontal probe
Plaque Index (PI) | 21 days
  Presence or absence of visible plaque evaluated with a periodontal probe
Plaque Index (PI) | 90 days
  Presence or absence of visible plaque evaluated with a periodontal probe
Gingival index (GI) | Baseline
  Presence or absence of changes in gingiva color
Gingival index (GI) | 7 days
  Presence or absence of changes in gingiva color
Gingival index (GI) | 21 days
  Presence or absence of changes in gingiva color
Gingival index (GI) | 90 days
  Presence or absence of changes in gingiva color
Periodontal pocket depth (PD) | Baseline
  Depth in millimeters with a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) at six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual), excluding third molar
Periodontal pocket depth (PD) | 90 days
  Depth in millimeters with a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) at six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual), excluding third molar
Clinical attachment level (CAL) | Baseline
  Depth in millimeters with a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) at six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual), except the third molar. Distance in millimeters from the cementoenamel limit to the bottom of the sulcus/periodontal pocket.
Clinical attachment level (CAL) | 90 days
  Depth in millimeters with a North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) at six sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual), except the third molar. Distance in millimeters from the cementoenamel limit to the bottom of the sulcus/periodontal pocket.
Bleeding on probing (BOP) | Baseline
  Presence of bleeding at the examined site up to 10 seconds after the examination.
Bleeding on probing (BOP) | 90 days
  Presence of bleeding at the examined site up to 10 seconds after the examination.
Microbiological evaluation | Baseline
  Real-time PCR with absolute quantification to confirm the number of colony-forming units (CFU) of bacterial samples from the six sites with the highest PD; specifically P gingivalis, T denticola, T forsythia, E nodatum and A. actinomycetemcomitans
Microbiological evaluation | 7 days
  Real-time PCR with absolute quantification to confirm the number of colony-forming units (CFU) of bacterial samples from the six sites with the highest PD; specifically P gingivalis, T denticola, T forsythia, E nodatum and A. actinomycetemcomitans
Microbiological evaluation | 21 days
  Real-time PCR with absolute quantification to confirm the number of colony-forming units (CFU) of bacterial samples from the six sites with the highest PD; specifically P gingivalis, T denticola, T forsythia, E nodatum and A. actinomycetemcomitans
Microbiological evaluation | 90 days
  Real-time PCR with absolute quantification to confirm the number of colony-forming units (CFU) of bacterial samples from the six sites with the highest PD; specifically P gingivalis, T denticola, T forsythia, E nodatum and A. actinomycetemcomitans

SECONDARY OUTCOMES:
Adverse effects | 7 days
  A survey was carried out on each participant at 7 and 21 days of the study to identify clinical adverse effects such as burning sensation, burning or pain in the oral mucosa, sensation of dryness or dryness, and changes in the perception of taste or the color in the teeth.
Adverse effects | 21 days
  A survey was carried out on each participant at 7 and 21 days of the study to identify clinical adverse effects such as burning sensation, burning or pain in the oral mucosa, sensation of dryness or dryness, and changes in the perception of taste or the color in the teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Plata, DDS MSc, Principal Investigator — Universidad El Bosque; Gloria Lafaurie, DDS MSc, Study Director — Unit of Basic Oral Investigation (UIBO) - Universidad El Bosque; David Díaz-Báez, DDS MSc, Principal Investigator — Unit of Basic Oral Investigation (UIBO) - Universidad El Bosque
Locations (1):
- Universidad El Bosque, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo DM, Castillo Y, Delgadillo NA, Neuta Y, Jola J, Calderon JL, Lafaurie GI. Viability and Effects on Bacterial Proteins by Oral Rinses with Hypochlorous Acid as Active Ingredient. Braz Dent J. 2015 Oct;26(5):519-24. doi: 10.1590/0103-6440201300388. PMID 26647939
- [Background] Lafaurie GI, Zaror C, Diaz-Baez D, Castillo DM, De Avila J, Trujillo TG, Calderon-Mendoza J. Evaluation of substantivity of hypochlorous acid as an antiplaque agent: A randomized controlled trial. Int J Dent Hyg. 2018 Nov;16(4):527-534. doi: 10.1111/idh.12342. Epub 2018 Apr 2. PMID 29608039